CLINICAL TRIAL: NCT06855641
Title: Patient Preference for Intraoperative Opioid Use and Early Recovery Following Non-Cardiac Surgery: Protocol for a Randomized Factorial Design Trial of Opioid-Free vs Opioid-Based Anesthesia (PERFECT TRIAL)
Brief Title: Effect of Patient Preference for Intraoperative Opioid Use on Early Postoperative Quality of Recovery
Acronym: PERFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Alexandre P. Joosten, Associate Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-24-5789
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-03

CONDITIONS: Opioid Analgesia; Quality of Recovery (QoR-15); Outcome Assessment; Opioid Free Anesthesia
Keywords: opioids; quality of recovery; analgesia; moderate risk surgery; postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The PERFECT trial is an interventional, pragmatic, partially randomized trial with factorial design.
Who Masked: Outcomes Assessor
Masking Description: quality of recovery will be done by research coordinators and research students ( undergraduate students) not involved in patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient choose his analgesia type (Experimental): The patient here can decide which type of analgesia he/she wants ( OFA vs OBA)
  Interventions: Procedure: Opioid based Anesthesia; Procedure: opioid free anesthesia
- Patient does not choose his analgesia strategy (Active Comparator): If the patient does not choose his analgesia strategy, he/she will be randomized to OFA or OBA
  Interventions: Procedure: Opioid based Anesthesia; Procedure: opioid free anesthesia

INTERVENTIONS:
Procedure: Opioid based Anesthesia — in this group, patient will receive standard of care at UCLA including fentanyl administration during surgery
Procedure: opioid free anesthesia — In this group, patients will not receive any opioids intraoperatively

SUMMARY:
Substituting the administration of opioids with a combination of alternative analgesics, known as opioid-free anesthesia (OFA), is gaining in popularity today and is typically administered as part of a larger multimodal strategy. However, OFA adoption is not as common today as one could expect from the potential benefits of limiting opioid use and patient involvement in the decision may impact its adoption. Relevant shared decision-making process with patients concerning the use or limited use of opioids could improve patient autonomy and empowerment. There have been no studies that have evaluated patient preference regarding opioid use and its potential impact on the quality of recovery.

The aim of this study is to compare the effect of patient preference on intraoperative opioid use on early postoperative quality of recovery following moderate risk laparoscopic/robotic abdominal surgery.

DETAILED DESCRIPTION:
Although opioid analgesic drugs are commonly used to relieve pain associated with surgery, they are not consequence free. Respiratory depression, postoperative nausea and vomiting (PONV), impaired gastrointestinal function, urinary retention are frequent concerns associated with their use. Moreover, the United States and many western countries are currently experiencing a significant health problem with opioid addiction and deaths due to overdose. Some opioid addiction pathways can trace their origin back to when a patient was first admitted to a hospital and received opioids in the setting of acute pain or surgery. As a result of this, there is likely a potential iatrogenic component to the current opioid abuse epidemic. Questioning the role of opioids is part of enhanced recovery after surgery programs, and good practice to reduce the risk of developing addiction and other side effects. Substituting the administration of opioids with a combination of alternative analgesics, known as opioid-free anesthesia (OFA), is gaining in popularity today and is typically administered as part of a larger multimodal strategy. However, OFA adoption is not as common today as one could expect from the potential benefits of limiting opioid use and patient involvement in the decision may impact its adoption. Relevant shared decision-making process with patients concerning the use or limited use of opioids could improve patient autonomy and empowerment. There have been no studies that have evaluated patient preference regarding opioid use and its potential impact on the quality of recovery.

The aim of this study is to compare the effect of patient preference on intraoperative opioid use on early postoperative quality of recovery following moderate risk laparoscopic/robotic abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Undergoing elective intermediate risk surgery under general anesthesia (robotic or laparoscopic assisted urological, gynecological or abdominal surgery).
* American Society Anesthesiologists physical status classification system grades of I-IV.
* English speaking.
* Informed consent signed.

Exclusion Criteria:

* Diagnosis of chronic pain
* Preoperative prescribed opioids
* Pregnancy or lactation.
* History of mental disorders.
* Contraindications to study drug (lidocaine, magnesium, dexmedetomidine, ketamine)
* Patient is participating in another interventional trial
* Patient is under judicial protection or is an adult under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Quality of recovery (QoR15) | Postoperative day 1
  The primary outcome will be the comparison of early postoperative quality of recovery (QoR) on postoperative day 1 (POD#1) using the validated QoR-15 score (as a whole, and each item separately) between patients who choose vs don't choose their anesthesia strategies. The minimum score is 0 and the maximum score is 150. The higher score, the better quality of recovery

SECONDARY OUTCOMES:
Quality of Recovery at postoperative day 2 | Postoperative day 2
  QoR15 at postoperative day 2 (same as the primary outcome but assessed at POD#2). The minimum score is 0 and the maximum score is 150. The higher score, the better quality of recovery
PONV incidence | Postoperative day 2
  Incidence of postoperative nausea and vomiting defined as the use in percentage of any antiemetic drug in the post-anesthesia care unit (PACU) and from PACU discharge to home discharge (usually between postoperative day 1 and 2)
Anesthesia satisfaction | Postoperative day 1
  Anesthesia satisfaction assessment with the Bauer questionnaire. Overall satisfaction and satisfaction by category prevalence (%). Self assessment. It contains 5 questions with 4 categories of answers (very satisfy- satisfy- dissatisfy - very dissatisfy). The proportion of each questions will be compared between groups
Postoperative opioid consumption | Postoperative 30
  opioid consumption in morphine equivalent (mg) from PACU arrival to hospital discharge and from hospital discharge to 30 days post-surgery
Intraoperative bradycardia | during surgery
  bradycardia incidence during surgery: defined as a heart rate < 40 per min with concomitant atropine administration (%)
Postoperative hypoxemia incidence | Postoperative day 2
  hypoxemia incidence defined as therapeutic oxygen supplementation to maintain SpO2 > 95% from PACU arrival to postoperative day 2
Health quality of life | Postoperative day 30
  Health quality of life on POD#30 with EuroQol5 dimension. Five-level version (EQ-5D-5L score) with visual analogic scale (for each question, you should answer among 5 propositions). The higher score, the better the quality of life of the patient.
Early quality of recovery on POD#1 | Postoperative day 1
  QoR15 at POD#1 depending on OFA vs OBA, whatever patient preferences. The minimum score is 0 and the maximum score is 150. The higher score, the better quality of recovery

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre JOOSTEN, MD PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Ronald Reagan medical center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gricourt Y, Boulos NM, Delaporte A, Alexander B, Besada S, Bakhit R, Toukhtarian A, Neuman I, Pearce D, Nourian MM, Chebishian A, Zhou A, Boktor J, Mayanja D, Grogan T, Boldt D, Cannesson M, Forget P, Joosten A. Patient preference for intraoperative opioid use and early recovery after noncardiac surgery: protocol for a randomised factorial design trial of opioid-free versus opioid-based anaesthesia (the PERFECT trial). BJA Open. 2025 Jun 18;15:100420. doi: 10.1016/j.bjao.2025.100420. eCollection 2025 Sep. PMID 40607110